CLINICAL TRIAL: NCT04732039
Title: Daily Life Activities in Patients Treated With Continuous-Flow Left Ventricular Assist Device
Brief Title: Daily Life Activities in Patients Treated With Continuous-Flow Left Ventricular Assist Devices
Acronym: Act-VAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Finn Gustafsson, Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: H-20049568
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Left Ventricular Failure, Unspecified
Keywords: left ventricular assist device; oxygen uptake; daily life activity; quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomized crossover study:
  1. Peak oxygen uptake vs VO2 measure during specific daily life activities in LVAD recipients
  2. Peak oxygen uptake vs VO2 measure during specific daily life activities in healthy controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LVAD recipients (Experimental): Peak oxygen uptake vs VO2 measure during specific daily life activities in LVAD recipients
  Interventions: Other: Measurement of peak oxygen uptake
- Healthy controls (Experimental): Peak oxygen uptake vs VO2 measure during specific daily life activities in healthy controls.
  Interventions: Other: Measurement of peak oxygen uptake

INTERVENTIONS:
Other: Measurement of peak oxygen uptake — Oxygen uptake measured on bike (pVO2) and during the conduction of specific daily life activities (ADL-VO2).

SUMMARY:
Investigation of oxygen uptake during daily life activities in HF patients with and without LVADs.

DETAILED DESCRIPTION:
In patients with terminal HF the gold standard for treatment is heart transplantation, though the Worldwide shortage of donor organs has led to increased use of implantable mechanical circulatory support devices. The treatment with implantable pumps in the form of a Continuous Flow Left Ventricular Assist Device (CF-LVAD, or simply LVAD) is extremely effective for a selected patient groups leading to significant improvement in survival and quality of life.

The device is a battery-powered flow pump that carries the blood from the left ventricle to the main artery, via a cannula, and thus relieves the failing left ventricle with up to 10 liters of blood per minute. An LVAD can be used both as lifelong support therapy (Destination Therapy, DT) or until transplantation can take place (Bridge therapy).

As patients today live for more than 10 years with the device as DT, the focus has shifted from mere survival to quality of life and physical ability.

In recent years, our research group showed that the pump speed and the patient's baseline heart rhythm (sinus rhythm vs atrial fibrillation) and reduced ability to regulate the intrinsic rhythm after implantation (chronotropic incompetence) are significant contributors to the reduced exercise capacity seen in this patient group.

Until now, studies have elucidated the work capacity of this patient group using a 6-minute walk test or bicycle test - none of these reflect how well the patient actually functions in his everyday life.

In this study, we will describe oxygen uptake related to specific daily activities (ADL-VO2) and compare these with the well-known maximum work capacity (percentage of expected oxygen uptake / pVO2) in this patient group.

ELIGIBILITY:
LVADs:

Inclusion Criteria:

* Implanted durable left ventricular assist device
* Age>18yrs
* Signed informed consent

Exclusion Criteria:

* No consent
* Not able to complete VO2 test (physicians decision)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
VO2 | Stable LVAD recipients on average 2 years after the implantation
  Oxygen uptake

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD,PhD,DMSci, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, DK, Denmark